CLINICAL TRIAL: NCT02800083
Title: A Multisite Randomized, Double-Blind, Placebo-Controlled Trial Evaluating Pitolisant (BF2.649) For Alcohol Use Disorder Treatment
Brief Title: A Trial Evaluating Pitolisant (BF2.649) in Alcohol Use Disorder Treatment
Acronym: PoC Alcohol
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Bioprojet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P15-14/BF2.649
Record Dates: First submitted 2016-06-07; First posted 2016-06-15 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-06

CONDITIONS: Alcohol Abuse, Nervous System
MeSH Terms: conditions — Alcohol-Induced Disorders, Nervous System | interventions — pitolisant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pitolisant (BF2.649) (Experimental): Histamine H3 receptor H3R antagonist/ inverse agonist
  Interventions: Drug: Pitolisant (BF2.649)
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pitolisant (BF2.649)
  Arms: Pitolisant (BF2.649)
Drug: Placebo
  Arms: Placebo

SUMMARY:
* The study primary end point is the decrease in the number of monthly heavy drinking days (HDD) (≥ 60 g/day in men and ≥ 40 g/d in women) from baseline to the end of the double blind Randomized Treatment (RT).
* The Secondary end points will be designed to assess safety and tolerability and to further investigate the effect of pitolisant on other alcohol use criteria (e.g. total alcohol consumption, number of abstinence days), craving as well as the improvement in mental health (depression, sleep) and quality of life.

  * Total alcohol consumption (TAC) from baseline to end of treatment. TAC was defined as mean daily alcohol consumption in g/day over a month (28 days).
  * Percent of patients without HDDs during the 24 weeks RT phase of the study. (Continuous Controlled Drinking=CCD)
  * Percent of Abstinent Days during RT phase (PAD)
  * Continuous Abstinence Duration from baseline during 24 weeks RT phase (CAD)
  * 4-week point prevalence abstinence at end of treatment
  * Improvement in alcohol biomarkers (e.g. ALAT, ASAT, % CDT) during 24 week RT phase
  * Craving (Obsessive Compulsive Drinking Scale) during 24 week RT phase
  * Beck Depression Inventory (BDI) during 24 week RT phase
  * Quality of sleep (Pittsburgh Sleep Quality Index) during RT phase.
  * Treatment retention during 24 week RT
  * Quality of life (SF-12) during RT phase
  * Percent patients without HDDs during the OL follow up period
  * Quality of life (SF-12) during OL phase
  * Quality of sleep (Pittsburgh Sleep Quality Index) during OL phase
  * Treatment retention OL phase Safety will be assessed by evaluation of treatment emergent adverse events (TEAE), physical examinations, clinical laboratory tests (blood chemistry, hematology, and urinalysis), subsequent end of treatment potential withdrawal, evaluation scales and physical examination, measurement of heart rate, blood pressure, and body weight at each study visit )V0-FU5). If at ECG Fridericia's corrected QT interval ≥ 500 ms or if difference to baseline is ≥ 60 ms it will be required to check ECG by second measurement after lying down 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with moderate or severe DSM-5 alcohol use disorder (based on the alcohol use disorders section of the MINI Plus)
* Ages 18-65.
* Low to moderate alcohol withdrawal symptoms: CIWA-Ar scale <10 at baseline assessment
* Normal weight: 18 kg/m2 ≤ BMI ≤ 35 kg/m2.
* Excessive alcohol use: number of heavy drinking days (≥ 60 g/day in men and ≥ 40 g/d in women) ≥15 during 30 days prior to screening and ≥7 during the 2 weeks between screening and baseline.
* Treatment-seeking, treatment goal: reduced drinking or abstinence
* If fertile, both males and females must agree to use effective birth control. Females of child-bearing potential must use a medically accepted effective method of birth control, agree to continue this method for the duration of the study and be negative to serum pregnancy test performed at the screening visit. Females should not be breast-feeding.
* Adequate social support according to the investigator to comply with the study requirements described in the protocol (e.g. transportation to and from trial site, self-rating scales, drug compliance, scheduled visits, etc.).
* Voluntarily expressed willingness to participate in the study, understanding protocol procedures and having signed and dated an informed consent prior to the start of protocol required procedures while not intoxicated (BAC<0.05).
* Willing to receive psychosocial support

Exclusion Criteria:

* History of delirium tremens, epilepsy, or withdrawal seizures
* Clinical depression or suicidality: Beck Depression Inventory (BDI) < 16 and suicidality (Item G =0)
* Recent illicit drug use, i.e. cannabis, cocaine, amphetamines or opioids.
* Clinically significant cardiovascular, hematologic, severe hepatic impairment or (FLTs> 3 ULN), renal (Stage 2 and 3 according to international classification of renal kidney disease), neurological, endocrinological abnormalities or abnormal clinical laboratory results (in most cases > 3ULN).
* History of serious head trauma or injury causing loss of consciousness that lasted more than 3 minutes.
* HIV positive; HCV positive; HBsAg positive
* History of psychosis, or current severe psychiatric disorder, e.g. schizophrenia, bipolar disorder, severe depression or organic brain syndrome unrelated to alcohol abuse
* Physical dependence on sedatives or hypnotics that requires pharmacologically supported detox.
* Receiving ongoing alcohol use disorder medication (e.g. Baclofen)
* Other active clinically significant illness, which could interfere with the study conduct or counter-indicate the study treatments or place the patient at risk during the trial or compromise the study participation.
* Known history of syncope, arrhythmia, myocardial infarction or any known significant ECG abnormality
* Known hypersensitivity to the tested treatment including active substance and excipients.
* Participation in clinical trial and receipt of investigational drug(s) during previous 60 days, except as explicitly approved by the Principal Investigator.
* Insufficient medical insurance according to local regulations.
* Pregnant woman or a pregnancy detected with a positive serum pregnancy test performed at the screening visit or lactating women
* Male subject who wants to conceive a child during the duration of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Monthly Heavy Drinking Days (HDD/month) | Change from Baseline of Monthly Heavy Drinking Days and at week 24

SECONDARY OUTCOMES:
Total daily Alcohol Consumption (TAC) | at week 24 versus Baseline
Percent of Abstinent Days during 24 weeks medication phase (PAD) | at week 24 versus Baseline
Improvement in alcohol biomarkers (ALAT, ASAT, % CDT) | at baseline , at week 4 , at week 8, at week 12, at week 16, at week 20 and at week 24. versus Baseline
Continuous Abstinence Duration during 24 weeks medication phase (CAD) | at week 24 versus Baseline
Obsessive Compulsive Drinking Scale (OCDC) | at week 24 versus Baseline
Time Line Follow Back (TLFB) | at week 24 versus Baseline
Alcohol Use Disorders Identification Test (AUDIT) | at week 24 versus Baseline
Pittsburgh Sleep Quality Index (PSQI) | at week 24 versus Baseline
Quality of Life (SF-12) | at week 24 versus Baseline